CLINICAL TRIAL: NCT00679211
Title: A Phase II, Single-Arm, Open-Label Study of Trastuzumab-Mcc-DM1 Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer
Brief Title: A Study of Trastuzumab-Mcc-DM1 Administered Intravenously to Patients With HER2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM4374g
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2013-05

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-positive breast cancer; HER2; MBC; Trastuzumab emtansine
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (1):
- Trastuzumab emtansine (Experimental): Trastuzumab emtansine (T-DM1) was administered to participants at a dose of 3.6 mg/kg by intravenous (IV) infusion every 3 weeks until documented disease progression, unmanageable toxicity, or study termination.
  Interventions: Drug: Trastuzumab emtansine [Kadcyla]

INTERVENTIONS:
Drug: Trastuzumab emtansine [Kadcyla] — Intravenous repeating dose
  Other Names: Trastuzumab-MCC-DM1; T-DM1

SUMMARY:
Study of trastuzumab emtansine (T-DM1) administered to patients with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed study-specific Informed Consent Form(s)
* Age ≥ 18 years
* Histologically documented breast cancer
* HER2-positive disease
* Metastatic breast cancer
* Disease progression on the last chemotherapy regimen received in the metastatic setting
* Prior treatment with an anthracycline, trastuzumab, a taxane, lapatinib, and capecitabine in the neoadjuvant, adjuvant, locally advanced, or metastatic setting and prior treatment with at least two lines of therapy (a line of therapy can be a combination of two agents or single-agent chemotherapy) in the metastatic setting
* At least two lines of anti-HER2 therapy must have been given in the metastatic setting as monotherapy or combined with chemotherapy or hormonal therapy. The HER2-targeted agent can include trastuzumab, lapatinib, or an investigational agent with HER2-inhibitory activity.
* A minimum of 6 weeks of trastuzumab for the treatment of metastatic disease is required
* Patients must have had at least 14 days of exposure in the metastatic setting to lapatinib and capecitabine (given together or separately) unless they were intolerant of lapatinib and/or capecitabine

Exclusion Criteria:

* Chemotherapy ≤ 21 days before enrollment
* Trastuzumab ≤ 21 days before enrollment
* Hormone therapy ≤ 7 days before enrollment
* Granulocyte-stimulating agent < 14 days before enrollment
* Investigational therapy ≤ 28 days before enrollment
* Previous radiotherapy for treatment of metastatic breast cancer ≤ 21 days before enrollment
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery, or other therapy to control symptoms from brain metastases within 3 months of the first study treatment
* History of intolerance (including Grade 3-4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
* History of exposure to the following cumulative doses of anthracyclines: Doxorubicin or liposomal doxorubicin > 500 mg/m^2; Epirubicin > 900 mg/m^2; Mitoxantrone > 120 mg/m^2 and idarubicin > 90 mg/m^2
* Peripheral neuropathy of Grade ≥ 3 per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
* History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma
* Current unstable angina
* History of symptomatic congestive heart failure (CHF), or ventricular arrhythmia requiring treatment
* History of myocardial infarction within 6 months of enrollment
* Left ventricular ejection fraction (LVEF) < 50% within 28 days of enrollment
* History of decreased LVEF to < 50% or symptomatic CHF with previous adjuvant trastuzumab treatment
* Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
* Current pregnancy or lactation
* Current known infection with human immunodeficiency virus (HIV), active hepatitis B, and/or hepatitis C virus
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Guardino, M.D., PhD., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between 13 August 2008 and 2 April 2009, 110 patients from 44 study sites in the United States were enrolled and treated in the study.
Period: Overall Study
Arm/Group | Trastuzumab Emtansine
Started | 110
Completed | 0
Not Completed | 110
Not completed — Progressive disease | 82
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 5
Not completed — Refused to undergo protocol procedures | 1
Not completed — Transferred to extension study TDM4529g | 12
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.1) [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response as Assessed Through Independent Radiologic Review
Description: Objective response was defined as a complete response (CR) or partial response (PR) determined on two consecutive occasions ≥ 4 weeks apart, assessed using Response Evaluation Criteria in Solid Tumors (RECIST).
  CR: the disappearance of all target lesions and all nontarget lesions and normalization of tumor marker level and no new lesions.
  PR: disappearance of all target lesions and persistence of ≥ 1 nontarget lesion(s) and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing nontarget lesions.
  The primary data cut-off date was 17 September 2009 (approximately 6 months after the last patient was enrolled). The final efficacy analysis was performed using a data cut-off date of 1 January 2010 (approximately 9 months after the last patient was enrolled).
Time Frame: From randomization until the primary analysis data cut-off date of September 2009 (6 months after last patient enrolled) and until the final efficacy analysis cut-off date of 1 January 2010 (approximately 9 months after the last patient enrolled).
Population: Treated population (patients who received at least one dose of T-DM1). Participants without a post-baseline tumor assessment were considered to be non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 6 Months of Follow-up; 9 Months of Follow-up: Trastuzumab emtansine (T-DM1) was administered to participants at a dose of 3.6 mg/kg by intravenous (IV) infusion every 3 weeks until documented disease progression, unmanageable toxicity, or study termination.
Arm/Group | 6 Months of Follow-up | 9 Months of Follow-up
Number analyzed (Participants) | 110 | 110
percentage of participants | 32.7 [24.1 to 42.1] | 32.7 [24.1 to 42.1]

2. Secondary Outcome: Duration of Objective Response as Assessed Through Independent Radiologic Review
Description: For participants who achieved an objective response, duration of objective response was defined as the time from the first tumor assessment that supported a participant's objective response to the time of disease progression or death on study (i.e., death from any cause within 30 days of the last dose of study drug), whichever occurred first. Response was assessed by the independent review facility.
  Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions.
  For participants who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate the duration of objective response.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Participants with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 36
months | NA [4.6 to NA] — The median duration of objective response was not reached due to a low number of events (defined as disease progression or death from any cause on study, whichever occurred first).

3. Secondary Outcome: Progression-free Survival as Assessed Through Independent Radiologic Review
Description: Progression-Free Survival (PFS) was defined as the time from the first day of study treatment to documented disease progression or death on study (i.e., death from any cause within 30 days of the last dose of study drug), whichever occurred first.
  Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Disease progression was assessed by the independent review facility.
  For patients who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Treated population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
months | 6.9 [4.2 to 9.5]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit Based on Independent Radiologic Review
Description: Clinical benefit was defined as participants who achieved an objective response (confirmed complete or partial response) between randomization and 1 January 2010, or with stable disease at 6 months. Stable disease at 6 months was defined as participants who achieved at least stable disease based on tumor assessments by the independent review facility, and remained alive and progression-free at 6 months.
  Stable disease was defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started, and no new lesions and/or unequivocal progression of existing nontarget lesions. Response was assessed by the independent review facility.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Treated population. Participants without a post-baseline tumor assessment were considered to have experienced no clinical benefit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
percentage of participants | 48.2 [38.8 to 57.9]

5. Secondary Outcome: Objective Response Based on Investigator Assessment
Description: Objective response was defined as a complete response (CR) or partial response (PR) determined on two consecutive occasions ≥ 4 weeks apart, assessed using Response Evaluation Criteria in Solid Tumors (RECIST). Response was assessed by the study Investigator.
  CR: the disappearance of all target lesions and all nontarget lesions and normalization of tumor marker level and no new lesions.
  PR: disappearance of all target lesions and persistence of ≥ 1 nontarget lesion(s) and/or the maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diameter of target lesions, and no new lesions or unequivocal progression of existing nontarget lesions.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Treated population. Participants without a post-baseline tumor assessment were considered to be non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
percentage of participants | 32.7 [24.1 to 42.1]

6. Secondary Outcome: Progression-free Survival Based on Investigator Assessment
Description: Progression-Free Survival (PFS) was defined as the time from the first day of study treatment to documented disease progression or death on study (i.e., death from any cause within 30 days of the last dose of study drug), whichever occurred first.
  Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions.
  For patients who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate PFS.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
months | 5.5 [4.1 to 7.5]

7. Secondary Outcome: Duration of Objective Response Based on Investigator Assessment
Description: For participants who achieved an objective response, duration of objective response was defined as the time from the first tumor assessment that supported a participant's objective response to the time of disease progression or death on study (i.e., death from any cause within 30 days of the last dose of study drug), whichever occurred first. Response was determined by the Investigator's assessment.
  Disease progression was at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions or the appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions.
  For participants who experienced no disease progression and did not die while on study, data were censored at the date of the last tumor assessment. Kaplan-Meier methodology was used to estimate the duration of objective response.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Participants with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 36
months | 9.7 [6.6 to NA] — Upper limit of the confidence interval not reached due to low number of events (defined as disease progression or death from any cause on study, whichever occurred first).

8. Secondary Outcome: Percentage of Participants With Clinical Benefit Based on Investigator Assessment
Description: Clinical benefit was defined as participants with an objective response (confirmed complete or partial response) or stable disease at 6 months. Patients with stable disease at 6 months were defined as patients who achieved at least stable disease based on tumor assessments and remained alive and progression free at 6 months. Response was based on the Investigator's assessment.
Time Frame: From randomization until 1 January 2010, approximately 9 months after the last participant was enrolled.
Population: Treated population. Patients without a post-baseline tumor assessment were considered to have experienced no clinical benefit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 110
percentage of participants | 46.4 [37.1 to 56.1]

ADVERSE EVENTS:
Time Frame: From the date of first dose until 26 April 2011, approximately 25 months of follow-up.
Arm/Group | Trastuzumab Emtansine
Serious Adverse Events (participants affected / at risk) | 29/110
Other Adverse Events (participants affected / at risk) | 105/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=110)
Atrial fibrillation (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Axillary pain (General disorders) | 2
Chest pain (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Bacteraemia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Blood culture positive (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Central nervous system necrosis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Influenza like illness (General disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Emtansine (N=110)
Thrombocytopenia (Blood and lymphatic system disorders) | 37
Anaemia (Blood and lymphatic system disorders) | 23
Leukopenia (Blood and lymphatic system disorders) | 6
Lacrimation increased (Eye disorders) | 9
Vision blurred (Eye disorders) | 7
Nausea (Gastrointestinal disorders) | 41
Constipation (Gastrointestinal disorders) | 27
Dry mouth (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 18
Diarrhoea (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 69
Pyrexia (General disorders) | 24
Chills (General disorders) | 11
Oedema peripheral (General disorders) | 11
Pain (General disorders) | 10
Chest pain (General disorders) | 7
Influenza like illness (General disorders) | 6
Urinary tract infection (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 15
Aspartate aminotransferase increased (Investigations) | 30
Alanine aminotransferase increased (Investigations) | 16
Blood alkaline phosphatase increased (Investigations) | 12
Weight decreased (Investigations) | 12
Blood lactate dehydrogenase increase (Investigations) | 10
Platelet count decreased (Investigations) | 8
Haemoglobin decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 25
Decreased appetite (Metabolism and nutrition disorders) | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Headache (Nervous system disorders) | 26
Neuropathy peripheral (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 7
Depression (Psychiatric disorders) | 11
Anxiety (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 7
Breast pain (Reproductive system and breast disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 9
Hot flush (Vascular disorders) | 7
Lymphoedema (Vascular disorders) | 7
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.